CLINICAL TRIAL: NCT02851342
Title: Graph-theoretical Analysis of Magnetoencephalographic Recordings as a Biomarker for Cognitive Deterioration in Multiple Sclerosis
Brief Title: GTA-MEG as a Biomarker for Cognition in MS
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: BRUMEG
Record Dates: First submitted 2016-07-25; First posted 2016-08-01 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis
Keywords: Cognition; MEG
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MS: patients with multiple sclerosis
- CO: matched control subjects

SUMMARY:
In this study, 100 persons with Multiple Sclerosis and 50 matched controls will be examined with magnetoencephalography (MEG), magnetic resonance imaging (MRI) and cognitive tests. The primary hypothesis for the study is: Interhemispheric connectivity, determined using graph theoretic analysis (GTA) on source-reconstructed MEG data, is a biomarker for cognitive deterioration in MS, which has value at the individual patient level.

DETAILED DESCRIPTION:
Procedures

Clinical assessment

* Disease type (Progressive onset/Relapsing onset)
* Disease phase (onset, relapsing remitting, secondary progressive, …)
* EDSS measurement (standard in the neurological examination)
* Time since last relapse (important for the exclusion criteria)
* Medication
* Level of education
* Pre-morbid Intelligence Quotient (IQ)

Symbol Digit Modalities Test (SDMT) - screening

* General
* In the final design of this study, the investigators will screen our patient group using the Symbol Digit Modalities Test (SDMT), a fast (5 min) and easy test that has been shown to be predictive of general cognitive impairment in MS probably due to the importance of information processing speed in cognitive deterioration in MS.
* This screening procedure will allow us to include an 'enriched' sample of MS patients; i.e. including patients with different cognitive abilities will allow us to assess correlations between brain network organization and cognition over a broader range of cognitive abilities.

MEG/EEG assessment

* General
* The subjects are asked to come to the MEG unit in the Université libre de Bruxelles (ULB) Erasmus Hospital in Anderlecht
* MEG measurements will be obtained using a Neuromag-306 Vector View system (Elekta). This scanner has 306 channels: 102 pairs of orthogonal planar gradiometers and 102 magnetometers. To aid artifact detection, electrooculograms (EOG) and electrocardiograms (ECG) were also recorded. Sampling frequency is 1000 Hertz (HZ).
* Subjects will be monitored for excessive eye-blinks. Although methods as independent component analysis (ICA) can remove these artefacts to some extent, too many eye-blinks may render the subsequent analyses impossible.
* Preparing the subject for the MEG assessment takes about 45 min.
* The patient's head movement will be continuously monitored.
* Resting-state
* Eyes Open

  1. 10 min
  2. Subjects will be asked to pay attention to a fixation cross
* Eyes Closed

  1. 10 min
  2. Subjects will be asked not to fall asleep
* Adjusted SDMT
* In this experiment, the patients are shown a code that links the numbers 1-9 to a certain symbol. For each trial, they also see one example that links a number to a symbol and they are asked to press the LEFT button if they think the example conforms with the presented code and the RIGHT button if they think otherwise. Subjects will be given a maximum of 6 s for each decision to be made and response timings will be recorded. The code that is presented varies with every example. This computerized set up of the SDMT was kindly provided by prof. Rypma. There is a pause of 2s between every decoding task. A total of 256 stimuli are presented, half of which are correct. The design follows the design by Leavitt et al. very closely (except for variable the interstimulus interval- 4,8,12 s - that was fixed to 3s in this design. Depending on the speed at which the subjects answers, this paradigm is expected to last between 9 and 10 min.
* Practice trial

  1. The subjects are shown 10 trials and their response is monitored. In this step, the researcher checks if the subject understands the paradigm.
* Actual paradigm

  1. The patients will be shown 256 trials, 50 % of which are correct.
  2. The total time for this experiment (at a speed of 2s per decision is : 9 min).
  3. The subjects won't receive any feedback from this part.
* A small break of 10 minutes in order not to fatigue the subjects too much.
* Auditory P300 paradigm
* The subjects are asked to press a button when they hear a high-pitched tone among a series of standard tones. The interstimulus interval will randomly shift between 1 and 1.5 s.
* Practice trial

  1. Subjects will first hear the standard tone 10 times (1000 Hz)
  2. Subjects will hear the target (high-pitched, 1500 Hz) tone 2 times
  3. Subjects will hear the distractor tone (500 Hz) 2 times
  4. The interstimulus interval will be sampled from the same distribution as the interstimulus interval used in the actual test
  5. Patients are not asked to press any buttons in this part.
* Actual test

  1. The subjects will hear a series of 400 tones. The total test time is therefore 8m20.
* 80 % of the tones will be frequent tones
* 10 % of the tones will be target tones, for which the subjects are asked to press a button
* 10 % of the tones will be distractor tones. Subjects are asked not to press any button in case of these distractor tones.
* The subjects won't get any feedback on their performance
* N-back test
* In the N-back test, a subjects sees a series of numbers (1-4) and is asked to compare the current stimulus to the N'th previous stimulus. In the case of a zero-back experiment, the subjects are asked to press a button when they see a certain number (e.g. 2).
* The experiment is designed as follows. There are three conditions imposing different loads on working memory (0-,1- and 2-back tasks). Each block lasts 30 s and there are eight blocks for each condition. The total registration time is therefore 12 min. The experiment is designed in agreement with the literature.
* Before the actual experiment, there will be a small practice trial including the three blocks (0-, 1- and 2-back task). This lasts approximately 2 min.
* Possible confounders:
* General:

  1. These confounders are to be administered right after the MEG recordings.
  2. These confounders are important as they may influence the cognitive results obtained during the MEG.
* Depression (Beck Depression Inventory)
* Fatigue (Fatigue scale for Motor and Cognitive Functions, FSMC)
* Brief International Cognitive Assessment for MS (BICAMS)
* (2) MRI assessment
* The informed consent asks for permission to analyse the T1 and T2 image, two images included in the standard clinical protocol, in the data analysis for the study. Furthermore, we will acquire and analyse a diffusor tensor imaging (DTI) measurement and a resting-state functional MRI image.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis according to the modified McDonald criteria
* Expanded Disability Status Scale (EDSS) below 6.0
* Providing informed consent
* Age between 18 and 55 years

Exclusion Criteria:

• Major medical or psychiatric pathology that potentially influences cognition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2016-04; Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
MEG Contrasts of parameter estimates (COPE) | 0 to 1000 msec post stimulus
  Contrasts (first-level or group-level) of parameter estimates based on averaged measured magnetic activity.

CONTACTS AND LOCATIONS:
Locations (1):
- National MS Center Melsbroek, Melsbroek, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No